CLINICAL TRIAL: NCT01350180
Title: A Prospective Study Assessing the Predictive Value of TMPRSS2-ERG Gene Fusion and PTEN Deletion in High Risk Prostate Cancer Patients
Brief Title: Assessing DNA Changes in High Risk Prostate Cancer to Determine Prognosis
Status: Withdrawn | Type: Observational
Sponsor: Dr. Tamim Niazi (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Dr. Tamim Niazi, Radiation Oncologist, Sir Mortimer B. Davis - Jewish General Hospital
Organization: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Other Study IDs: MP-JGH-10-032
Record Dates: First submitted 2011-04-26; First posted 2011-05-09 (Estimated); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer
Keywords: biochemical failure; hormonal therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
One of the biggest problems facing prostate cancer patients and their treating physicians is who needs to be treated and when. Common clinical and pathological parameters are useful (PSA, Gleason score, etc.) but do not clearly predict who will benefit from treatment and who will fail. Genetic markers for tumor aggressivity would be of greater value. The finding that the TMPRSS2-ERG gene fusion is associated with an increase risk of cancer progression is important. TMPRSS2 is controlled by androgen (testosterone) and ERG is part of a family of proteins which have a role in controlling cell growth, cell specialization and producing tumors. As a consequence of this gene fusion, production of the ERG protein increases in the presence of testosterone and could be key to the development of prostate cancer, resistance to treatment and poor outcome. The PTEN gene is known to have a role as a tumor suppressor. Its deletion is a contributing factor in the development of prostate cancers and poor outcome. The coexistence of the two markers could be associated with a higher risk of recurrence.

To date there have been no studies regarding the presence of either of these two markers or their coexistence in high risk prostate cancer patients who, despite radiation therapy and androgen suppression, develop biochemical failure (their PSA levels rise once again). Patients participating in the PCS IV study (high risk prostate cancer treated with radiation therapy plus either 18 or 36 months of hormonal suppression) who have had biochemical failure or 3 years of follow-up post hormonal therapy will be approached.

Tumor blocks from consenting patients will be collected and analyzed for the presence of the TMPRSS2-ERG gene fusion and the PTEN deletion at the Pathology Department of the Jewish General Hospital. Statistical analysis will be carried out to see whether either or both markers are present, whether they are associated with certain clinical and pathological high risk factors, and whether they can be used to predict which patients will fail treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients with prostate cancer post radical radiation therapy and LHRH agonist treated in PCSIV clinical trial
* biochemical failure (PSA nadir + 2) or minimum follow-up of 3 years post completion of hormonal therapy
* high risk group

  1. gleason score 8-10
  2. PSA ≥ 20 ng/ml
  3. T3 or T4

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: high risk prostate cancer patients having received radical radiation and hormonal therapy in either biochemical failure or 3-year post end of hormonal therapy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
number of patients with biochemical failure showing the TMPRSS2-ERG gene fusion and/or PTEN deletion | recruitment over 2 years
  biopsy samples of patients treated for high risk prostate cancer with radical radiation and hormonal therapy who have either biochemical failure or 3-year post treatment follow-up free of cancer recurrences will be tested for the TMPRSS2-ERG gene fusion and the PTEN deletion. The results between the two groups will be compared to see if either DNA changes are an indicator of disease recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Tamim Niazi, MD, Principal Investigator — Sir Mortimer B. Davis - Jewish General Hospital
Locations (8):
- Canada (8):
  - Hôpital de Gatineau, Gatineau, Quebec
  - CHUM-Notre- Dame, Montreal, Quebec
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - CHUQ, L'Hôtel-Dieu de Québec, Québec, Quebec
  - CHUS - Hôpital Fleurimont - Sherbrooke, Sherbrooke, Quebec
  - Centre Hospitalier régional de Trois-Rivières, Trois-Rivières, Quebec